CLINICAL TRIAL: NCT02377700
Title: Initial Safety and Performance of the COR-VP-001 Vascular Patch in Pediatric Patients Undergoing Bidirectional Cava-pulmonary Anastomosis
Brief Title: Safety and Performance of a Vascular Patch in Pediatric Patients Undergoing Bidirectional Cava-pulmonary Anastomosis
Acronym: XEL-CR-06
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xeltis (Industry)
Collaborators: Q-Med Scandinavia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XEL-CR-06
Record Dates: First submitted 2015-02-18; First posted 2015-03-03 (Estimated); Results first posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Heart Defects, Congenital
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Xeltis Vascular Patch, Model COR-VP-001 (Experimental): Patients implanted with the vascular patch during staged bidirectional cava-pulmonary anastomosis.
  Interventions: Device: Xeltis Vascular Patch, Model COR-VP-001

INTERVENTIONS:
Device: Xeltis Vascular Patch, Model COR-VP-001 — The intended use of the Xeltis Vascular Patch, Model COR-VP-001 is to augment pulmonary artery and thereby improve hemodynamics by increasing blood flow to the lungs in patients with congenital pulmonary artery obstructions as an initial part of the staged procedure of a bidirectional cava-pulmonary anastomosis

SUMMARY:
Xeltis developed biodegradable patch prosthesis, the Vascular Patch Model COR-VP-001, to be used as a vascular patch to augment the pulmonary trunk and pulmonary arteries. The prosthesis is immediately mechanically functional, while its physiochemical characteristics should enable cell infiltration and tissue formation.

The Xeltis Vascular Graft Model COR-VP-001 is specifically designed to improve surgical outcomes by reducing synthetic material related complications and improving hemodynamic characteristics.

DETAILED DESCRIPTION:
Xeltis has developed a medical device for treating pediatric cardiovascular patients requiring RVOT reconstruction. Xeltis' mission is to offer 'Solutions for a Lifetime' to cardiovascular patients. Xeltis has developed a unique technology based on novel biodegradable bio-materials allowing the regrowth of natural heart valves or blood vessels in patients' bodies from their own cells.

The principle of Xeltis' COR technology (COR stands for Cardiovascular Organ Regeneration) is to implant a biodegradable prosthesis of a blood vessels that is shaped like the part to be replaced. The prosthesis is immediately mechanically functional, while its physiochemical characteristics should enable cell infiltration and tissue formation. Tissue is regenerated and functional by the time the polymer is biodegraded.

ELIGIBILITY:
Inclusion Criteria:

1. Patient requiring a bidirectional cava-pulmonary anastomosis
2. Male or Female
3. Age: 2 months to 16 years

Exclusion Criteria:

1. Main Exclusion Criteria Arrhythmias as determined by ECG and/or at the investigator's discretion
2. Other clinically significant malformations
3. Coagulation disorders as defined by INR outside its normal value, PTT >ULN and Fibrinogen <LLN and/or at the investigator's discretion
4. HIV-infection
5. Syphilis (Treponema pallidum)
6. Hepatitis-B and/or -C virus infection
7. Unwillingness of Parental/legal guardian to give consent
8. Treatment with other investigational products
9. Known or suspected noncompliance, drug or alcohol abuse of the parents/legal guardian
10. Inability of the parents/legal guardian to follow the procedures of the study, e.g. due to language problems
11. Participation of the patient in another study within 30 days preceding and during the present study
12. Previous enrolment of the patient into the current study
13. Enrolment of the investigator's family members, employees and other dependent persons

Ages: 2 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2014-06; Primary Completion 2015-09 (Actual); Study Completion 2020-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leo Bockeria, Professor, Principal Investigator — Bakoulev Center for Cardiovascular Surgery
Locations (1):
- Bakoulev Center for Cardiovascular Surgery, Moscow, Russia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Xeltis Vascular Patch, Model COR-VP-001
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Xeltis Vascular Patch, Model COR-VP-001
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 3.9 [0.5 to 16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Region of Enrollment [Number; unit: participants]
  Russia | 5

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patch Related Serious Adverse Events.
Description: Evaluation of the safety of the COR-VP-001 as defined by number of patients having patch related post-operative complications requiring surgery, intervention or leading to death up to 12 months post implantation
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Xeltis Vascular Patch, Model COR-VP-001
Number analyzed (Participants) | 5
Participants | 0

2. Secondary Outcome: Number of Subjects With Loss of Functionality of the Patch.
Description: Evaluation of the performance of the COR-VP-001 by analyzing the incidence of loss of functionality requiring intervention within up to 12 months post implantation.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Xeltis Vascular Patch, Model COR-VP-001
Number analyzed (Participants) | 5
Participants | 0

3. Secondary Outcome: Histological Evaluation
Description: Number of patients with histological evaluation of the patch material obtained during the planned reoperation within up to 12 months after implantation
Time Frame: up to 12 Months after Implant
Measure: Count of Participants; unit: Participants
Arm/Group | Xeltis Vascular Patch, Model COR-VP-001
Number analyzed (Participants) | 5
Participants | 1

ADVERSE EVENTS:
Arm/Group | Xeltis Vascular Patch, Model COR-VP-001
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xeltis Vascular Patch, Model COR-VP-001 (N=5)
Stenosis in the bi-directional cava pulmonary anastomosis (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xeltis Vascular Patch, Model COR-VP-001 (N=5)
Sick sinus syndrome and bundle branch block (Cardiac disorders) | 1 (1)
Supraventricular tachycardia and atrial fibrillation (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No